CLINICAL TRIAL: NCT02077452
Title: A Randomized, Double-blinded, Placebo-Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Ascending Doses of HMS5552 in Adult Patients With Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HMS5552 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hua Medicine Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HMM0102
Record Dates: First submitted 2014-03-02; First posted 2014-03-04 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glucokinase activator; Phase I; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Dorzagliatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- HMS5552 dose 1 (Experimental): HMS5552 25~400mg. Oral administration, twice per day.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 2 (Experimental): HMS5552 25~400mg. Oral administration, twice per day.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 3 (Experimental): HMS5552 25~400mg. Oral administration, twice per day.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 4 (Experimental): HMS5552 25~400mg. Oral administration, once per day.
  Interventions: Drug: HMS5552; Drug: Placebo
- HMS5552 dose 5 (Experimental): HMS5552 25~400mg. Oral administration, twice per day.
  Interventions: Drug: HMS5552; Drug: Placebo

INTERVENTIONS:
Drug: HMS5552
Drug: Placebo

SUMMARY:
The objectives of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of HMS5552 following multiple ascending doses in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This will be a randomized, double-blind and placebo-controlled study with multiple oral doses of HMS5552 given to patients with type 2 diabetes mellitus who never accepted anti-diabetic drug for treatment before.

The primary objective is to characterize the safety and tolerability of HMS5552 following multiple ascending doses in patients with type 2 diabetes mellitus after BID dosing for 8 days.

The secondary objectives include:

1. To determine the single dose and steady state pharmacokinetics of HMS5552 in patients with type 2 diabetes
2. To evaluate the single dose and steady state pharmacodynamics of HMS5552 in patients with type 2 diabetes
3. To further explore food-effect on HMS5552 pharmacokinetics and pharmacodynamics

A maximum total of 80 patients (10 in each dose group and assuming a maximum of 5~8 dose levels). There will be 8 active and 2 placebo patients in each dose group. The safety, tolerability, pharmacokinetics and pharmacodynamics data after each dose cohort will be reviewed in blinded fashion before escalation to the next dose cohort.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with type 2 diabetes
* Age: 18 to 65 years
* BMI: 20 to 29 kg/m2
* Mentally, physically and legally eligible to give informed consent.
* Willingness to adhere to the protocol requirement.

Exclusion Criteria:

* Subjects with type 1 diabetes
* Episodes of hypoglycemia
* Unstable cardiovascular diseases
* Hepatic diseases
* Kidney disease
* Mental or central nervous system diseases
* Clinical abnormal findings in ECG, labs and physical exams

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of HMS5552 will be assessed by adverse event monitoring, physical examinations, 12 lead ECGs, vital sign, and safety laboratory measurements. | up to 15 days after study drug administration

SECONDARY OUTCOMES:
The single dose and steady state pharmacokinetics (with food and fasting) of HMS5552 will be described by estimating parameters of AUCinf, AUC0-t, Cmax, Tmax, Ae, T1/2, CL/f, CLr/f, accumulation index and fluctuation index. | up to day 8 post-dose
  1. Single dose (Day 1) plasma and urine pharmacokinetic parameters (postprandial)
  2. Single dose (Day 3) plasma and urine pharmacokinetic parameters (fasting)
  3. Steady state (Day 7) plasma and urine pharmacokinetic parameters (postprandial)
  4. Steady state (Day 8) plasma and urine pharmacokinetic parameters (fasting)
The single dose and steady state (fasting and postprandial) pharmacodynamic variables will include maximum absolute and percent change in plasma glucose level, AUC0-4, AUC0-16, AUC16-24, AUC0-24 hr of plasma glucose. | up to 4 hour post-dose and up to 24 hour post-dose
Insulin, C-peptide, glucagon and glucagon-like peptide 1 up to 6hr post-dose following single dose and steady state (fasting and postprandial) | up to 6 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dalong ZHU, MD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School